CLINICAL TRIAL: NCT02460471
Title: Palliative Radiotherapy for Advanced Head and Neck Carcinomas, a Phase II Study
Brief Title: Palliative Radiotherapy Protocol in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Bernard Fortin MD MSc FRCPC, principal investigator, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11020
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Neoplasms; Quality of Life
Keywords: Radiotherapy; Palliative Care; IMRT
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- palliative radiation therapy (Experimental): 25 Gy in 5 daily fractions
  Interventions: Radiation: palliative radiation therapy

INTERVENTIONS:
Radiation: palliative radiation therapy — thermoplastic mask immobilization. CT in treatment position. radiation dose of 25 Gy in 5 daily fractions over one week 6 MV photons by intensity modulation. Target volume is the symptomatic tumour volume with a 5 mm margin

SUMMARY:
Phase II prospective study or Palliative Radiotherapy of 25 Gy in 5 fractions, Intensity Modulated, for frail patients with incurable head and neck cancer. Comprehensive Quality of life (QLQ-C30, head and neck module, QLQ C15 PAL) and toxicity data (CTCAE v 4.0) collected.

DETAILED DESCRIPTION:
Patients deemed too frail for radical treatment or incurable because of tumour extension, as determined by an experienced tumour board, were eligible for this study of palliative radiotherapy delivered by intensity modulation, 25 Gy in 5 daily fractions over one week. This study was conducted in two academic centers.

ELIGIBILITY:
Inclusion Criteria:

* Able to give an informed consent
* Able to complete QOL questionnaires
* Deemed incurable by an experienced tumour board or unwilling to receive a radical course of radiation therapy
* Presence of measurable disease
* Biopsy proven squamous or salivary cancer of the head and neck region
* Expected survival of at least 2 months.

Exclusion Criteria:

* Pregnancy
* No previous RT to the neck and no plan to receive concomitant chemotherapy
* Special histology (Lymphoma, small cell cancer, metastasis from a site other than the head and neck region)
* Unavailable for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Quality of life | from radiation treatment until 24 months planned follow-up or death
  EORTC QLQ-C30 questionnaire (QLQ-C15-PAL and H&N35 modules)

SECONDARY OUTCOMES:
Toxicity (CTCAE v 4.0 graded) | from radiation treatment until 24 months planned follow-up or death
  CTCAE v 4.0 graded toxicities

OTHER OUTCOMES:
Progression free survival | from radiation treatment until 24 months planned follow-up or progression or death
Overall survival | from radiation treatment until 24 months planned follow-up or death

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Fortin, MD MSc, Principal Investigator — Maisonneuve Rosemont Hospital, University of Montreal
Locations (2):
- Canada (2):
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

REFERENCES:
- [Derived] Fortin B, Khaouam N, Filion E, Nguyen-Tan PF, Bujold A, Lambert L. Palliative Radiation Therapy for Advanced Head and Neck Carcinomas: A Phase 2 Study. Int J Radiat Oncol Biol Phys. 2016 Jun 1;95(2):647-53. doi: 10.1016/j.ijrobp.2016.01.039. Epub 2016 Jan 28. PMID 27020111